CLINICAL TRIAL: NCT01980563
Title: Optimizing Ovarian Stimulation for IVF and ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2010/367
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Efficiency in Terms of Mature Oocyte Yield
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasound (Active Comparator)
  Interventions: Procedure: ultrasound; Procedure: combined monitoring
- combined monitoring (Active Comparator)
  Interventions: Procedure: ultrasound; Procedure: combined monitoring

INTERVENTIONS:
Procedure: ultrasound
Procedure: combined monitoring

SUMMARY:
Monitoring ovarian stimulation for in vitro fertilization (IVF) and intracytoplasmatic sperm injection (ICSI) can be simplified by reducing the procedure to measuring follicles by ultrasound. Proponents of a simplified procedure claim that the procedure can be reduced to simple monitoring by ultrasound while maintaining results (numbers of mature oocytes, percentage of pregnancy and live birth rates). On the other hand simultaneous blood sampling for measuring hormone levels is still the state of the art in many clinics. A large review (Cochrane review) stated that "although there was no clear evidence for a better outcome, combined cycle monitoring was still recommended until it could be proven that ovarian hyperstimulation can be avoided without hormonal monitoring". Investigators therefore perform a study that compares the results between 2 groups: those with ultrasound monitoring and those with combined monitoring. Deciding when to plan the retrieval of the oocytes can depend on subtle differences in the number of large follicles measured by ultrasound, but also on hormonal levels in the blood of the patient. Therefore the investigators planned a randomized study in the group of patients with combined monitoring. The investigators examined if delaying the moment for planning the moment of oocyte retrieval by 24 hours had any effect on the number of mature oocytes and pregnancy rates and what the effect of rising progesterone levels might be. The investigators hypothesis was that combined monitoring could lead to better results since recent studies have thought that rising progesterone levels, if found, have a negative impact on pregnancy rates. On the other hand the investigators expect to find that waiting for larger follicles in cases with normal progesterone levels lead to a better oocyte yield.

ELIGIBILITY:
inclusion criteria:

* absence of ovarian cysts
* both ovaries present

exclusion criteria:

* ovarian cysts
* not both ovaries present

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 416 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The number of mature oocytes obtained. | 1 day

SECONDARY OUTCOMES:
The number of fertilized oocytes/good quality embryos | at the moment of egg retrieval up to embryo transfer, assessed up to 100 months
Pregnancy rate | 12 months after egg retrieval
clinical pregnancy rate | 12 months after egg retrieval
ongoing pregnancy rate | 12 months after egg retrieval
live birth rate for each individual transferred embryo | 12 months after egg retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vandekerckhove, MD, Principal Investigator — Fertility clinic
Locations (1):
- University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Vandekerckhove F, Gerris J, Vansteelandt S, De Baerdemaeker A, Tilleman K, De Sutter P. Delaying the oocyte maturation trigger by one day leads to a higher metaphase II oocyte yield in IVF/ICSI: a randomised controlled trial. Reprod Biol Endocrinol. 2014 Apr 23;12:31. doi: 10.1186/1477-7827-12-31. PMID 24758641